CLINICAL TRIAL: NCT03521570
Title: Phase II Study of IMRT Re-Irradiation With Concurrent/Adjuvant Nivolumab in Patients With Locoregionally Recurrent or Second Primary Squamous Cell Cancer of the Head and Neck
Brief Title: Intensity-Modulated Radiation Therapy & Nivolumab for Recurrent or Second Primary Head & Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); The Cleveland Clinic (Other); Medical College of Wisconsin (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nabil F. Saba, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00100923; NCI-2018-00064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4221-17 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, IMRT) (Experimental): Patients receive nivolumab IV over 30 minutes on weeks -2, 0, 2, 4, and 6 and undergo IMRT once daily beginning on week 0 for up to 6-6.5 weeks. Beginning week 10, patients receive nivolumab IV over 30 minutes every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: IMRT; Biological: Nivolumab

INTERVENTIONS:
Radiation: IMRT — Undergo intensity-modulated radiation therapy
  Other Names: Intensity-Modulated Radiation Therapy; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well intensity-modulated radiotherapy and nivolumab work together in treating patients with head and neck squamous cell cancer that has come back. Intensity-modulation radiation therapy uses varying intensities of radiation beams to kill cancer cells and shrink tumors, thereby reducing the damage to nearby healthy tissue. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Giving intensity-modulated radiation therapy and nivolumab may work better at treating head and neck squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the 1-year progression-free survival (PFS) for patients with recurrent or second primary head and neck squamous cancer treated with intensity-modulated radiation therapy (IMRT) re-irradiation with concurrent and adjuvant nivolumab.

SECONDARY OBJECTIVES:

I. Evaluate the 1-year (yr) overall survival (OS) of patients treated with re-irradiation and nivolumab.

II. Evaluate patient quality of life (QOL).

III. Evaluate patterns of failure including local, regional and distant failure rates at 1 yr.

IV. Identify and estimate the incidence rate of acute and late toxicities associated with combined re-irradiation and concurrent and adjuvant nivolumab.

TERTIARY OBJECTIVE:

I. To identify potential biomarkers related to clinical benefit to concurrent and adjuvant nivolumab and re-irradiation in patients with recurrent or second primary (RSP) head and neck squamous cell carcinoma (HNSCC).

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on weeks -2, 0, 2, 4, and 6 and undergo IMRT once daily beginning on week 0 for up to 6-6.5 weeks. Beginning week 10, patients receive nivolumab IV over 30 minutes every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years from the beginning of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent squamous cell carcinoma or a second primary arising in a previously irradiated field
* Life expectancy of greater than 6 months
* Patients cannot have distant metastases and have to be candidates for curative re-irradiation
* Patients with salivary gland tumors are excluded (patients with nasopharynx or sinonasal cancers can participate)
* Patients with unresectable disease are eligible
* Patients who undergo surgical resection will be allowed regardless of human papilloma virus (HPV) status provided they have one of the following criteria:

  * Positive margins on pathology
  * Evidence of extracapsular spread on nodal pathology
  * Gross residual disease on postoperative or simulation imaging
  * N2/3 disease
  * T3/4 disease
  * Multifocal perineural invasion and/or lymphovascular space invasion
* The majority of the anticipated target volume (> 50%) must have been previously treated to ≥ 40 Gy; prior radiation therapy (RT) must have been completed > 6 months prior to initiation of IMRT reirradiation; if previous RT records are unavailable, investigators can estimate the dose to previously treated tissues based on completion notes or other treatment history
* An Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Granulocytes > 1500/mm³
* Platelets > 100,000/mm³
* Bilirubin < 1.5 mg/dl
* Creatinine < 1.5 mg/dl
* No other concurrent invasive malignancies treated for the past year (localized prostate cancer or early stage skin cancer are not exclusion criteria)
* Patients with carotid artery involvement or encasement will be allowed provided they have no symptoms related to carotid involvement
* No prior exposure to immunotherapy agents
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any known factors that would pose a contraindication to receiving nivolumab
* Recursive partitioning analysis (RPA) class III patients defined as those expected to begin reirradiation within 2 years of first course of radiation therapy AND are percutaneous endoscopic gastrostomy (PEG) dependent or have a tracheostomy (patients who have undergone total laryngectomy are not excluded)
* Patients with metastases
* Prior treatment with a programmed cell death protein-1 (PD-1)/programmed death-ligand 1 (PD-L1) inhibitor
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment
* Patients with primary salivary gland cancers are excluded
* Patients who have had chemotherapy or biological therapy within 4 weeks of registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disease requiring systemic steroids, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or breast-feeding
* Patients with known active human immunodeficiency virus (HIV), hepatitis (hep) B, or hep C infection
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F. Saba, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Saba NF, Wong SJ, Nasti T, McCook-Veal AA, McDonald MW, Stokes WA, Anderson AM, Ekpenyong A, Rupji M, Abousaud M, Rudra S, Bates JE, Remick JS, Joshi NP, Woody NM, Awan M, Geiger JL, Shreenivas A, Samsa J, Ward MC, Schmitt NC, Patel MR, Higgins KA, Teng Y, Steuer CE, Shin DM, Liu Y, Ahmed R, Koyfman SA. Intensity-Modulated Reirradiation Therapy With Nivolumab in Recurrent or Second Primary Head and Neck Squamous Cell Carcinoma: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jul 1;10(7):896-904. doi: 10.1001/jamaoncol.2024.1143. PMID 38780927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab, IMRT)
Started | 62
Completed | 51
Not Completed | 11
Not completed — Not eligible | 11

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 20
Age, Continuous [Mean (Full Range); unit: years] | 62 [56 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 39
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-Free Survival (PFS)
Description: 95% confidence interval will be estimated by Kaplan-Meier method for all participants.
Time Frame: 1 year from study start
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
Participants | 27

2. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Will be assessed using Kaplan-Meier method.
Time Frame: 1 year from study start
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
percentage of participants | 84.4 [74.4 to 95.7]

3. Secondary Outcome: Number of Participants With Pattern of Failure
Description: To evaluate patterns of failure as local, regional, or distant.
Time Frame: 1 year from study start
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
Participants | 2

4. Secondary Outcome: Number of Participants With Incidence of Acute Adverse Events
Description: Acute toxicities will be identified and their incidence rate estimated.
Time Frame: Up to 1 year from study start
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
percentage of participants
  fatigue | 82.4
  dermatitis | 58.8
  dysphagia | 54.9
  mucositis | 49
  dry mouth | 47.1
  Lymphopenia | 11.8

5. Secondary Outcome: Number of Participants With Incidence of Late Adverse Events
Description: Late toxicities will be identified and their incidence rate estimated.
Time Frame: 2 years from study start
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
Participants | 3

6. Secondary Outcome: Quality of Life (QOL)
Description: The FACT-HN (Functional Assessment of Cancer Therapy-Head and Neck) (version 4) consists of a cancer-specific questionnaire, FACT-G (Functional Assessment of Cancer Therapy - General), in addition to 12 H&N cancer-specific items (the HN subscale).The Functional Assessment of Cancer Therapy-Head and Neck Quality of Life questionnaire may be completed by the patient using paper or electronically. FACT-HN total score ranges between 0 and 148. The higher the score, the better the QOL
Time Frame: At baseline, end of Intensity-Modulated Radiation Therapy, and weeks 18, 30, 52, and 104, baseline and month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Nivolumab, IMRT)
Number analyzed (Participants) | 51
score on a scale
  Baseline | 68 (89.2)
  End of IMRT | 62.5 (90)
  Week 18 | 62 (93.4)
  Week 30 | 74.6 (101)
  Week 52 | 59 (94.5)
  Week 104 | 59 (94.5)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Nivolumab, IMRT)
All-Cause Mortality (participants affected / at risk) | 24/51
Serious Adverse Events (participants affected / at risk) | 24/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab, IMRT) (N=51)
Death (General disorders) | 24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab, IMRT) (N=51)
Oral pain (Gastrointestinal disorders) | 12
Mucositis oral (Gastrointestinal disorders) | 24
Constipation (Gastrointestinal disorders) | 17
Agitation (Psychiatric disorders) | 3
Dysphagia (Gastrointestinal disorders) | 28
Dermatitis radiation (Injury, poisoning and procedural complications) | 30
Anorexia (Metabolism and nutrition disorders) | 20
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 40
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperthyroidism (Endocrine disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 24
Peripheral sensory neuropathy (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 12
Insomnia (Psychiatric disorders) | 8
Diarrhea (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 28
Dysgeusia (Nervous system disorders) | 21
Anal hemorrhage (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Chills (General disorders) | 4
Oral dysesthesia (General disorders) | 1
Weight loss (Investigations) | 11
Lymphocyte count decreased (Investigations) | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Depression (Psychiatric disorders) | 10
Creatinine increased (Investigations) | 5
Pain (General disorders) | 11
Vaginal infection (Infections and infestations) | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1
Dysesthesia (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Esophageal pain (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 13
Vomiting (Gastrointestinal disorders) | 4
Bronchial infection (Infections and infestations) | 1
Oral dysesthesia (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 8
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6
Hypothyroidism (Endocrine disorders) | 14
Lymphedema (Vascular disorders) | 5
Colitis (Gastrointestinal disorders) | 3
Mucosal infection (Infections and infestations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 7
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 4
Memory impairment (Nervous system disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Alkaline phosphatase increased (Investigations) | 2
Paresthesia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 7
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Aspartate aminotransferase increased (Investigations) | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 12
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6
Hearing impaired (Ear and labyrinth disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 2
Eye pain (Eye disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 5
Facial pain (General disorders) | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 7
Facial nerve disorder (Nervous system disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Infective myositis (Infections and infestations) | 1
Myasthenia gravis (Nervous system disorders) | 1
White blood cell decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Eyelid function disorder (Eye disorders) | 1
Edema face (General disorders) | 4
Dysphasia (Nervous system disorders) | 1
Sinusitis (Infections and infestations) | 3
Heart failure (Cardiac disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Tremor (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 2
Weight gain (Investigations) | 2
Platelet count decreased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Neck edema (General disorders) | 4
Cataract (Eye disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Wound infection (Infections and infestations) | 1
Flu like symptoms (General disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Cardiac troponin I increased (Investigations) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Salivary duct inflammation (Gastrointestinal disorders) | 5
Ear pain (Ear and labyrinth disorders) | 5
Dizziness (Nervous system disorders) | 9
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Floaters (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Localized edema (General disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Stoma site infection (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 1
Dysarthria (Nervous system disorders) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2
Non-cardiac chest pain (General disorders) | 2
Malaise (General disorders) | 1
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1
Thrush (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 2
Edema limbs (General disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Skin infection (Infections and infestations) | 1
Obesity (Metabolism and nutrition disorders) | 1
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Blurred vision (Eye disorders) | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Stomach pain (Gastrointestinal disorders) | 1
Stomal ulcer (Injury, poisoning and procedural complications) | 1
Palpitations (Cardiac disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Flushing (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
Meningitis (Infections and infestations) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT03521570/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03521570/ICF_000.pdf